CLINICAL TRIAL: NCT04527250
Title: Comparison of the Pharmacokinetic Parameters of ASC41, a Randomized, Double-blind, Placebo-controlled in Healthy Subjects After Single and Multiple Doses
Brief Title: A Study of the Relative Bioavailability of ASC41 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASC-ASC41-I-CTP-02
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Experimental:1mg (Experimental): ASC41 one tablet (1mg) single oral dose at Day 1 and once daily for 14 days from Day 14 to Day 27.
  Interventions: Drug: ASC41
- Experimental:2mg (Experimental): ASC41 two tablets (2mg) single oral dose at Day 1 and two tablets daily for 14 days from Day 14 to Day 27.
  Interventions: Drug: ASC41
- Experimental:5mg (Experimental): ASC41 one tablet (5mg) single oral dose at Day 1 and once daily for 14 days from Day 14 to Day 27.
  Interventions: Drug: ASC41
- Experimental:10mg (Experimental): ASC41 two tablets (10mg) single oral dose at Day 1.
  Interventions: Drug: ASC41
- Experimental:20mg (Experimental): ASC41 four tablets (20mg) single oral dose at Day 1.
  Interventions: Drug: ASC41
- Placebo:1mg (Placebo Comparator): ASC41 placebo one tablet (1mg) single oral dose at Day 1 and once daily for 14 days from Day 14 to Day 27.
  Interventions: Drug: ASC41 placebo
- Placebo:2mg (Placebo Comparator): ASC41 placebo two tablets (2mg) single oral dose at Day 1 and two tablets daily for 14 days from Day 14 to Day 27.
  Interventions: Drug: ASC41 placebo
- Placebo:5mg (Placebo Comparator): ASC41 placebo one tablet (5mg) single oral dose at Day 1 and once daily for 14 days from Day 14 to Day 27.
  Interventions: Drug: ASC41 placebo
- Placebo:10mg (Placebo Comparator): ASC41 placebo two tablets (10mg) single oral dose at Day 1.
  Interventions: Drug: ASC41 placebo
- Placebo:20mg (Placebo Comparator): ASC41 placebo four tablets (20mg) single oral dose at Day 1.
  Interventions: Drug: ASC41 placebo

INTERVENTIONS:
Drug: ASC41 — ASC41,1mg/table;5mg/table
  Arms: Experimental:10mg; Experimental:1mg; Experimental:20mg; Experimental:2mg; Experimental:5mg
Drug: ASC41 placebo — ASC41 placebo,1mg/table;5mg/table
  Arms: Placebo:10mg; Placebo:1mg; Placebo:20mg; Placebo:2mg; Placebo:5mg

SUMMARY:
The objective of this study is to compare the pharmacokinetic parameters of ASC41 in healthy subjects after single and multiple oral dosing.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the tolerability, safety pharmacokinetics and pharmacodynamic (biomarkers) of ASC41 tables in a randomized, double-blind, placebo-controlled single- and multiple-dose phase I clinical trial in healthy subjects the study. The effects of ASC41 on LDL-C and other lipid parameters (TG, TC, HDL-C, etc.) will be observed after repeated administration of ASC41 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-45 (including boundary value). 2. Male weight ≥ 50kg, female weight ≥ 45kg;BMI ranges from 19 to 30kg/m2 (boundary value included).

  3. She is of childbearing potential and is non-pregnant and willing to use adequate contraception from screening (within 30days from the first administration)until one month after the End of Study visit.

  4. The pregnancy test of female subjects during the screening period is negative.

  5. During the screening period, fasting low-density lipoprotein cholesterol (110mg/dl < fasting (LDL-C) < 190mg/ dL.

  6. Those who voluntarily sign the informed consent.

Exclusion Criteria:

* 1. Patients with a history of thyroid disease or intolerance to beta blockers or abnormal thyroid function indicators during screening; 2. Previous history of fainting, fainting needle or fainting blood for unknown reasons.

  3. Previous liver disease, or ALT, ASL and direct bilirubin in screening period exceed the normal range.

  4. Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (HCV Ab), HIV antibody (HIV Ab) and syphilis antibody are tested positive.

  5. People who have taken special diet (including carambola, dragon fruit, mango, grapefruit, orange, etc.) or drunk alcohol, or had strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion within 2 weeks before taking the study drug.

  6. Heavy smokers (14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL spirits, or 100 mL wine;Smoking daily ≥ 5 sticks) and no smoking or alcohol prohibition during the study period.

  7. Ingesting chocolate, any food or drink containing caffeine or xanthine in the 24 hours prior to taking the study drug.

  8. Patients who had donated blood or lost blood of more than 400ml within 3 months before taking the study drug.

  9. Those who have participated in other clinical trials and received study drug treatment within 3 months before taking study drug.

  10. In addition to the above, the researchers judge that the participants are not suitable to participate in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of ASC41 in healthy volunteers | Up to 32 days
  Evaluation of the safety and tolerability of ASC41 in healthy volunteers

SECONDARY OUTCOMES:
Cmax of ASC41 | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 32 days.
  Evaluate the Peak Plasma Concentration after single and multiple oral doses of ASC41 administered to Chinese healthy volunteers.
Tmax of ASC41 | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 32 days.
  Evaluate the Time to reach the maximum plasma concentration after single and multiple oral doses of ASC41 administered to Chinese healthy volunteers.
AUC of ASC41 | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 32 days.
  Evaluate the Area under the plasma concentration versus time curve after single and multiple oral doses of ASC41 administered to Chinese healthy volunteers.
t1/2 of ASC41 | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 32 days.
  Evaluate the Terminal-Phase Half-Life after single and multiple oral doses of ASC41 administered to Chinese healthy volunteers volunteers.
CL/F of ASC41 | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 32 days.
  Evaluate the Apparent Systemic Clearance after single and multiple oral dose of ASC41 administered to Chinese healthy volunteers.
Vd/F of ASC41 | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 32 days.
  Evaluate the Apparent Volume of Distribution after single and multiple oral dose of ASC41 administered to Chinese healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan provincial people's hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided